CLINICAL TRIAL: NCT02904343
Title: Evaluation of Domestic Hemodialysis Machine (WEGO DBB-27C) : A Multi-center Clinical Study
Brief Title: Evaluation of Domestic Hemodialysis Machine: A Multi-center Clinical Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsors want to stop the study.
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xiangmei Chen, Professor,Chief physician,Academician of Chinese Academy of Engineering, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2015-046-01
Record Dates: First submitted 2016-08-22; First posted 2016-09-16 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Hemodialysis
Keywords: hemodialysis machine; quality; safety; domestic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of domestic hemodialysis machine (Experimental)
  Interventions: Device: domestic hemodialysis machine
- Group of imported hemodialysis machine (Active Comparator)
  Interventions: Device: imported hemodialysis machine

INTERVENTIONS:
Device: domestic hemodialysis machine — WEGO, DBB-27C
  Arms: Group of domestic hemodialysis machine
Device: imported hemodialysis machine — Fresenius, 4008s
  Arms: Group of imported hemodialysis machine

SUMMARY:
An important reason for the costs of hemodialysis treatment in China are expensive is the hemodialysis machine and related products mainly rely on imports. Hemodialysis machine is the basis equipment of the hemodialysis treatment. After years of research and development, China has had the domestic hemodialysis machine. However, due to the lack of control studies of domestic and imported hemodialysis machine, thus causing the domestic hemodialysis machine promotion has been hindered. The aim of this study is to verify the quality and safety of domestic hemodialysis machine.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18, male or female
2. Maintenance hemodialysis duration>3 months
3. Regular hemodialysis,3 times a week,4 hours per session
4. Sign the written informed consent

Exclusion Criteria:

1. Acute kidney injury
2. Prepare to transfer to kidney transplantation or peritoneal dialysis in a year.
3. Positive in Hepatitis B virus, hepatitis C virus, syphilis or HIV
4. Pregnancy or lactation
5. Under other drug trial
6. Acute infection, severe heart, lung, liver, nervous diseases, malignant tumor
7. Can not be treated in accordance with the research program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Adverse reactions associated with the use of dialysis machines | 0 to 3 months

SECONDARY OUTCOMES:
The results of endotoxin level of dialysate | 0,1,2,3 months
  endotoxin level of dialysis fluid at outlet
The results of bacterial culture of dialysate | 0,1,2,3 months
  bacterial culture of dialysis fluid at outlet
Clearance rate of uremic toxins | 0,1,2,3 months